CLINICAL TRIAL: NCT02225353
Title: A Randomized, Open-Label, Controlled, Multi-Center Study on the Efficacy of a Sustained Release Progesterone Cerclage Cervical Pessary at Doses of 6.3 g or 7.7 g for the Prevention of Preterm Birth and a Maximum Duration of 20 Weeks.
Brief Title: Efficacy Study of a Cervical Pessary Containing Progesterone for the Prevention of Preterm Delivery
Acronym: PCP002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC12012/10IEI-9339
Record Dates: First submitted 2014-08-04; First posted 2014-08-26 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Preterm Birth
Keywords: Preterm birth; Short cervix; Cervical Pessaries; Progesterone
MeSH Terms: conditions — Premature Birth | interventions — Progesterone; Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Progesterone Cervical Pessary 6.3 g (Experimental): 90 pregnant women with Progesterone Cervical Pessary
  Interventions: Drug: Progesterone Cervical Pessary 6.3 g
- Progesterone Cervical Pessary 7.7 g (Experimental): 90 pregnant women with Progesterone Cervical Pessary
  Interventions: Drug: Progesterone Cervical Pessary 7.7 g
- Progesterone 200 mg vaginal capsules (Active Comparator): 90 pregnant women using Progesterone 200 mg vaginal capsules daily
  Interventions: Drug: Progesterone 200 mg vaginal capsules

INTERVENTIONS:
Drug: Progesterone Cervical Pessary 6.3 g — Progesterone Cervical Pessary low dose
  Arms: Progesterone Cervical Pessary 6.3 g
Drug: Progesterone 200 mg vaginal capsules — Progesterone 200 mg vaginal capsules daily
  Other Names: Hormoral (Trade Mark) Capsules
  Arms: Progesterone 200 mg vaginal capsules
Drug: Progesterone Cervical Pessary 7.7 g — Progesterone Cervical Pessary high dose
  Arms: Progesterone Cervical Pessary 7.7 g

SUMMARY:
Assess the efficacy of 2 Cervical Pessaries containing 6.3 g and 7.7 g micronized progesterone for the prevention of preterm delivery, established through spontaneous birth before gestation weeks 32 (31 weeks and 6 days) and 34 (33 weeks and 6 days), when the pessary is inserted during weeks 16th and 24th and removed at 36 weeks and 6 days in pregnant women at high risk of premature birth.

DETAILED DESCRIPTION:
Participant selection will be performed by screening the general population of pregnant women with single fetus monitored by the Hospital Healthcare Network, to investigate by serial transvaginal ultrasound performed between gestation weeks 16 (0 day to 7 days) and 24 (0 day to 7 days) those patients who have a cervical length between 10 mm and 25 mm, and/or women with a single fetus and cervical length ≥10 mm presenting one or more of the following risk factors:

1. preterm birth prior to 35 (34 weeks and 6 days) weeks of gestation;
2. premature rupture of membranes prior to 35 (34 and 6 days) weeks of gestation.

After insertion of the pessary or beginning of the administration with vaginal progesterone capsules and until 28 weeks of gestation, participants in the 3 treatment groups will be monitored every 4 weeks at the most or more often, if the site has established so as a control standard. After 28 weeks, patients should be monitored every 2 weeks.

The proportions of spontaneous preterm delivery before gestation weeks 32 and 34 will be compared between the control group and the 2 groups with the pessaries containing different doses of progesterone.

ELIGIBILITY:
Inclusion Criteria:

* Women with a single pregnancy and a cervical length of 10 mm - 25 mm between 16 and 24 weeks of gestation, without any previous factors.
* Women with a single pregnancy with 10 mm or more cervical length between 16 and 24 weeks of gestation, and pre-existing risk factors risk factors for preterm birth:
* Previous preterm birth before week 35.
* Previous rupture of membranes before week 35

Exclusion Criteria:

* Pregnancies with:

  * Major fetal abnormalities, such as lethal malformations or malformations requiring pre- or post-natal surgery; and fetal death before inclusion into the study.
  * History of rupture of membranes or prophylactic cerclage before study entry.
* Cervical or vaginal injuries prior to insertion of the pessary (e.g., cervical erosion secondary to trauma, infection, or carcinoma; vesicovaginal or rectovaginal fistulas).
* Unconscious, severely ill or mentally disabled patients, or under 16 years of age.
* Patients for whom use of progesterone is contraindicated.
* Patients with history of thrombosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2013-09-02 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (4):
- Chile (4):
  - Universidad de Chile, Hospital Barros Luco, Santiago
  - Complejo Asistencial Dr. Sótero del Río (CASR), Santiago
  - Unidad de Alto Riesgo Obstétrico y Medicina Perinatal y en el Centro Perinatal Oriente (CERPO), Hospital Santiago Oriente, Dr. Luis Tisné Brousse, Santiago
  - Universidad de Chile, Hospital Clínico San Borja Arriarán, Santiago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dodd JM, Crowther CA, Cincotta R, Flenady V, Robinson JS. Progesterone supplementation for preventing preterm birth: a systematic review and meta-analysis. Acta Obstet Gynecol Scand. 2005 Jun;84(6):526-33. doi: 10.1111/j.0001-6349.2005.00835.x. PMID 15901258
- [Background] Berghella V. Novel developments on cervical length screening and progesterone for preventing preterm birth. BJOG. 2009 Jan;116(2):182-7. doi: 10.1111/j.1471-0528.2008.02008.x. PMID 19076950
- [Background] Jayasooriya GS, Lamont RF. The use of progesterone and other progestational agents to prevent spontaneous preterm labour and preterm birth. Expert Opin Pharmacother. 2009 Apr;10(6):1007-16. doi: 10.1517/14656560902851403. PMID 19351272
- [Background] Newcomer J. Pessaries for the treatment of incompetent cervix and premature delivery. Obstet Gynecol Surv. 2000 Jul;55(7):443-8. doi: 10.1097/00006254-200007000-00023. PMID 10885649
- [Background] Arabin B, Halbesma JR, Vork F, Hubener M, van Eyck J. Is treatment with vaginal pessaries an option in patients with a sonographically detected short cervix? J Perinat Med. 2003;31(2):122-33. doi: 10.1515/JPM.2003.017. PMID 12747228
- [Background] Goya M, Pratcorona L, Merced C, Rodo C, Valle L, Romero A, Juan M, Rodriguez A, Munoz B, Santacruz B, Bello-Munoz JC, Llurba E, Higueras T, Cabero L, Carreras E; Pesario Cervical para Evitar Prematuridad (PECEP) Trial Group. Cervical pessary in pregnant women with a short cervix (PECEP): an open-label randomised controlled trial. Lancet. 2012 May 12;379(9828):1800-6. doi: 10.1016/S0140-6736(12)60030-0. Epub 2012 Apr 3. PMID 22475493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial started on 02 Sep 2013 with the enrollment of the first participant and was completed on 13 Mar 2017 when the last participant completed the last follow-up examination according to the protocol. 271 participants signed and informed consent. All 271 were randomized and treated.
Groups:
- Progesterone Cervical Pessary (6.3 g); Progesterone Cervical Pessary (7.7 g): Cervical Pessary (PCP) with sustained release of progesterone. The PCP is inserted by investigator to participant at risk of preterm birth and remains installed with no further intervention except at the time of removal.
- Progesterone 200 mg Vaginal Capsules: Progesterone 200 mg vaginal capsules: Progesterone 200 mg vaginal capsules daily by participant.
Period: Overall Study
Arm/Group | Progesterone Cervical Pessary (6.3 g) | Progesterone Cervical Pessary (7.7 g) | Progesterone 200 mg Vaginal Capsules
Started | 91 | 90 | 90
Completed | 87 | 84 | 75
Not Completed | 4 | 6 | 15
Not completed — Lost to Follow-up | 0 | 1 | 3
Not completed — Protocol Violation | 4 | 5 | 12

BASELINE CHARACTERISTICS:
Population: Intent-to-treat.
Groups:
- Progesterone Cervical Pessary (6.3 g); Progesterone Cervical Pessary (7.7 g): Cervical pessary (PCP) with sustained release of progesterone. The PCP is inserted by investigator to participant (at risk of preterm birth) and remains installed with no further intervention except at the time of removal.
- Total: Total of all reporting groups
Arm/Group | Progesterone Cervical Pessary (6.3 g) | Progesterone Cervical Pessary (7.7 g) | Progesterone 200 mg Vaginal Capsules | Total
Number analyzed (Participants) | 91 | 90 | 90 | 271
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 91 | 90 | 90 | 271
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.57 (6.50) | 27.60 (6.20) | 28.18 (5.16) | 27.78 (5.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 90 | 90 | 271
  Male | NA — Male was an exclusion criterion | NA — Male was an exclusion criterion | NA — Male was an exclusion criterion | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 91 | 90 | 90 | 271
Region of Enrollment [Number; unit: participants]
  Chile | 91 | 90 | 90 | 271
Height [Mean (Standard Deviation); unit: meter] | 1.57 (0.06) | 1.58 (0.06) | 1.58 (0.05) | 1.58 (0.05)
Weight [Mean (Standard Deviation); unit: kilogram] | 66.65 (13.36) | 71.26 (14.06) | 70.62 (12.73) | 69.50 (13.50)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter] | 27.03 (4.92) | 28.61 (5.45) | 28.23 (4.56) | 27.95 (5.01)
Medical History - Prior Preterm Birth [Count of Participants; unit: Participants] | 55 | 55 | 50 | 160
Medical History - Prior Pregnancy Premature Rupture of Membrane [Count of Participants; unit: Participants] | 24 | 20 | 17 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Not Giving Birth Before Week 32 and Week 34 of Gestation
Description: To assess the efficacy of Cerclage Pessaries containing 6.3 g and 7.7 g micronized progesterone for the prevention of preterm delivery, established through spontaneous parturition before gestation weeks 32 (31 weeks and 6 days) and 34 (33 weeks and 6 days), when the pessary is inserted between weeks 16 and 24 and removed at 36 weeks and 6 days in pregnant women at high risk of premature delivery.
  For the purpose of this analysis, pregnancies were no longer considered as high risk for the event if delivery occurred at week 34 of gestation and beyond. Gestational age was determined by the last menstruation date and were confirmed by measurement of the craniocaudal length obtained in the first trimester ultrasound, or by measurement of the cephalic circumference in the second trimester ultrasound predominating the actual date of the last menstrual period.
  The number of participants not giving birth before 32 weeks and 34 weeks are reported.
Time Frame: Up to 36 weeks of gestational age
Population: 271 participants comprised the Intention-to-treat analysis (ITT) population at baseline, 268 participants at gestation week 32, and 262 participants at gestation week 34.
Measure: Count of Participants; unit: Participants
Groups:
- Progesterone Cervical Pessary (6.3 g): Cervical Pessary with sustained release of progesterone.Single placement and removal by investigator site.
- Progesterone Cervical Pessary (7.7 g): Cervical Pessary with sustained release of progesterone. Single placement and removal by investigator site.
Arm/Group | Progesterone Cervical Pessary (6.3 g) | Progesterone Cervical Pessary (7.7 g) | Progesterone 200 mg Vaginal Capsules
Number analyzed (Participants) | 91 | 90 | 90
Participants
  No birth before 32 weeks: number analyzed (Participants) | 90 | 90 | 88
  No birth before 32 weeks | 73 | 71 | 67
  No birth before 34 weeks: number analyzed (Participants) | 89 | 88 | 85
  No birth before 34 weeks | 66 | 64 | 61

2. Secondary Outcome: Number of Participants With Premature Rupture of Membranes
Description: A participant with premature rupture of membrane typically recalls a sudden gush of fluid loss from the vagina, or steady loss of small amounts of fluid. Participants who reported vaginal discharge were examined by a physician.
Time Frame: Up to 36 weeks of gestational age
Population: Intention-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Progesterone Cervical Pessary (6.3 g) | Progesterone Cervical Pessary (7.7 g) | Progesterone 200 mg Vaginal Capsules
Number analyzed (Participants) | 91 | 90 | 90
Participants | 1 | 4 | 3

3. Secondary Outcome: Anatomical Feature: Length of the Uterine Cervix
Description: During the pregnancy the length of the uterine cervix will be assessed. The rational is that premature birth is associated with uterine cervix shortening. The length of the cervix was determined using ultrasound examination. A positive change from baseline indicates a positive development, i.e. less likely to result in a preterm birth. The comparison between premature an normal birth initially planned by the protocol was not analyzed.
Time Frame: Up to 36 weeks of gestational age. Results are reported for all assessments from baseline through final visit, for a total of 8 visits, and for up to 36 weeks of gestational age.
Population: Intention-to-treat (ITT).
Measure: Mean (Standard Deviation); unit: millimeter
Groups:
- Progesterone Cervical Pessary (6.3 g); Progesterone Cervical Pessary (7.7 g): Cervical Pessary with sustained release of progesterone. Single placement and removal by investigator site.
Arm/Group | Progesterone Cervical Pessary (6.3 g) | Progesterone Cervical Pessary (7.7 g) | Progesterone 200 mg Vaginal Capsules
Number analyzed (Participants) | 91 | 90 | 90
millimeter
  Baseline Visit: number analyzed (Participants) | 91 | 89 | 89
  Baseline Visit | 28.69 (9.06) | 29.62 (8.66) | 28.44 (8.55)
  Visit 2: number analyzed (Participants) | 82 | 78 | 76
  Visit 2 | 28.51 (8.30) | 30.34 (7.63) | 29.29 (10.37)
  Visit 3: number analyzed (Participants) | 74 | 75 | 69
  Visit 3 | 27.54 (7.27) | 29.06 (7.65) | 30.76 (8.28)
  Visit 4: number analyzed (Participants) | 69 | 71 | 64
  Visit 4 | 27.82 (7.12) | 27.60 (7.91) | 29.37 (8.16)
  Visit 5: number analyzed (Participants) | 61 | 67 | 62
  Visit 5 | 27.53 (7.40) | 26.55 (7.81) | 28.63 (10.16)
  Visit 6: number analyzed (Participants) | 41 | 43 | 41
  Visit 6 | 27.42 (7.62) | 27.28 (9.36) | 27.49 (8.32)
  Visit 7: number analyzed (Participants) | 28 | 24 | 18
  Visit 7 | 30.43 (9.39) | 27.95 (8.85) | 28.83 (8.00)
  Final Visit: number analyzed (Participants) | 49 | 47 | 38
  Final Visit | 22.98 (8.06) | 25.07 (7.49) | 23.64 (9.26)

4. Secondary Outcome: Anatomical Feature: Position of the Uterine Cervix
Description: During the pregnancy the position of the uterine cervix will be assessed. The rational being that premature birth is associated with uterine cervix positioning. The position of the cervix was determined using transvaginal ultrasound examination. In the change from baseline visit a positive value change indicated that the investigator believed that the position of the cervix changed in a positive manner to facilitate a term birth. The comparison between premature an normal birth initially planned by the protocol was not analyzed. The results reported are the degrees of the cervix position relative to the longitudinal axis of the uterus.
Time Frame: as for outcome 3
Population: Intention-to-treat (ITT).
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Progesterone Cervical Pessary (6.3 g) | Progesterone Cervical Pessary (7.7 g) | Progesterone 200 mg Vaginal Capsules
Number analyzed (Participants) | 91 | 90 | 90
degrees
  Baseline Visit: number analyzed (Participants) | 54 | 58 | 40
  Baseline Visit | 114.54 (22.58) | 112.59 (22.48) | 112.85 (20.03)
  Visit 2: number analyzed (Participants) | 43 | 43 | 31
  Visit 2 | 111.47 (23.33) | 115.02 (19.56) | 109.74 (23.56)
  Visit 3: number analyzed (Participants) | 40 | 39 | 32
  Visit 3 | 110.81 (17.78) | 109.83 (25.65) | 115.36 (24.93)
  Visit 4: number analyzed (Participants) | 38 | 40 | 28
  Visit 4 | 105.58 (21.35) | 117.61 (18.63) | 113.29 (26.20)
  Visit 5: number analyzed (Participants) | 31 | 32 | 25
  Visit 5 | 108.99 (21.97) | 115.50 (19.15) | 113.26 (15.21)
  Visit 6: number analyzed (Participants) | 17 | 16 | 15
  Visit 6 | 112.96 (17.41) | 114.50 (21.61) | 121.65 (15.89)
  Visit 7: number analyzed (Participants) | 15 | 14 | 6
  Visit 7 | 118.93 (14.10) | 110.51 (20.94) | 124.37 (13.32)
  Final Visit: number analyzed (Participants) | 29 | 26 | 18
  Final Visit | 104.30 (23.98) | 113.42 (24.76) | 115.44 (16.14)

5. Secondary Outcome: Acceptability and Tolerance of Use of the Cerclage Pessary
Description: A questionnaire was planned to be used to compare acceptability and tolerance in the insertion, during pregnancy and during the extraction of Cerclage Pessary.
  Data from this questionnaire was not collected.
Time Frame: Up to 36 weeks of gestational age
Population: No participants were analyzed
Arm/Group | Progesterone Cervical Pessary (6.3 g) | Progesterone Cervical Pessary (7.7 g) | Progesterone 200 mg Vaginal Capsules
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Adverse Events Related With the Use of Treatment
Description: The number of adverse events reported were analyzed as being related with the treatment as well as for unexpectedness.
Time Frame: Up to 36 weeks of gestational age
Population: Intention-to-treat (ITT)
Measure: Number; unit: events
Units Other Than Participants: number of adverse events
Arm/Group | Progesterone Cervical Pessary (6.3 g) | Progesterone Cervical Pessary (7.7 g) | Progesterone 200 mg Vaginal Capsules
Number analyzed (Participants) | 91 | 90 | 90
Number analyzed (number of adverse events) | 200 | 248 | 200
events
  AE related to use of treatment | 31 | 22 | 2
  Unexpected serious adverse events | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: up to 36 weeks of gestational age (participants were in the trial for up to 20 weeks).
Description: Treatment emergent adverse events.
Groups:
- Progesterone Cervical Pessary 6.3 g: 91 pregnant women with Progesterone Cervical Pessary
  Progesterone Cervical Pessary: Progesterone Cervical Pessary: 6.3 g Progesterone Cervical Pessary: 7.7 g
- Progesterone Cervical Pessary 7.7 g: 90 pregnant women with Progesterone Cervical Pessary
  Progesterone Cervical Pessary: Progesterone Cervical Pessary: 6.3 g Progesterone Cervical Pessary: 7.7 g
Arm/Group | Progesterone Cervical Pessary 6.3 g | Progesterone Cervical Pessary 7.7 g | Progesterone 200 mg Vaginal Capsules
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/90 | 0/90
Serious Adverse Events (participants affected / at risk) | 36/91 | 35/90 | 33/90
Other Adverse Events (participants affected / at risk) | 77/91 | 73/90 | 65/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Progesterone Cervical Pessary 6.3 g (N=91) | Progesterone Cervical Pessary 7.7 g (N=90) | Progesterone 200 mg Vaginal Capsules (N=90)
Breast abscess (Infections and infestations) | 0 | 0 | 2
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 3
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 2
Hypertensive crisis (Vascular disorders) | 0 | 1 | 1
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 1
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 4 | 3
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Shortened cervix (Reproductive system and breast disorders) | 10 | 9 | 19
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 1 | 0 | 0
Cerebral ventricle dilatation (Nervous system disorders) | 1 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Polihidroamnios (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 3 | 0 | 0
Ventricular hypoplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Drug use disorder (Psychiatric disorders) | 1 | 0 | 0
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 0 | 4 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 2 | 0
Pelvic pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 1 | 0
Premature labor (Pregnancy, puerperium and perinatal conditions) | 17 | 6 | 2
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Bacteriuria (Infections and infestations) | 1 | 0 | 0
Foetal cerebrovascular disorder (Nervous system disorders) | 1 | 1 | 0
Vaginal erosion (Reproductive system and breast disorders) | 0 | 1 | 0
Multiple congenital anomalies (Congenital, familial and genetic disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Vaginal infection NOS (Reproductive system and breast disorders) | 1 | 0 | 0
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Coital bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Progesterone Cervical Pessary 6.3 g (N=91) | Progesterone Cervical Pessary 7.7 g (N=90) | Progesterone 200 mg Vaginal Capsules (N=90)
Anaemia (Blood and lymphatic system disorders) | 11 | 5 | 5
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Congenital uterine anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 3 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 4 | 2
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 3
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 3 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 7 | 2
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 3 | 1 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 14 | 5 | 2
Bronchitis (Infections and infestations) | 2 | 3 | 0
Cervicitis (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gastrenteritis (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 12 | 11 | 6
Vaginal infection (Infections and infestations) | 3 | 0 | 1
Vaginitis gardnerella (Infections and infestations) | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 11 | 7 | 8
Vulvovaginal candidasis (Infections and infestations) | 3 | 1 | 4
Vulvovaginitis (Infections and infestations) | 13 | 6 | 11
Tooth infection (Infections and infestations) | 0 | 0 | 1
Gynaecological chlamydia infection (Infections and infestations) | 0 | 1 | 0
Ureaplasma infection (Infections and infestations) | 2 | 2 | 2
Mycoplasma infection (Infections and infestations) | 0 | 2 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 16 | 11 | 10
Vaginitis chlamydial (Infections and infestations) | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Amniocentesis abnormal (Investigations) | 0 | 0 | 2
Ultrasound uterus (Investigations) | 1 | 1 | 0
Ultrasound uterus abnormal (Investigations) | 1 | 1 | 1
Ureaplasma test positive (Investigations) | 0 | 1 | 0
Mycoplasma test positive (Investigations) | 1 | 1 | 0
Foetal renal imaging abnormal (Investigations) | 0 | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 2
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pubic pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 6
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Facial paralysis (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 8 | 2 | 12
Tension headache (Nervous system disorders) | 0 | 0 | 1
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 6 | 11 | 7
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 3 | 4 | 2
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Uterine hypotonus (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 3
Umbilical cord abnormaility (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 11 | 12 | 9
Uterine contractions abnormal (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 1
Uterine irritability (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 12 | 6 | 11
Pruritus genital (Reproductive system and breast disorders) | 0 | 3 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 16 | 22 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 3 | 1
Vuvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 1
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 1 | 0
Genital discharge (Reproductive system and breast disorders) | 4 | 0 | 1
Vaginal erosion (Reproductive system and breast disorders) | 1 | 0 | 0
Cervix oedena (Reproductive system and breast disorders) | 1 | 0 | 0
Shortened cervix (Reproductive system and breast disorders) | 0 | 1 | 2
Vulvovaginal pain (Reproductive system and breast disorders) | 2 | 4 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Utricaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT02225353/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT02225353/SAP_001.pdf